CLINICAL TRIAL: NCT00063102
Title: A Phase II Study of ABT-751 in Patients With Breast Cancer Refractory to Taxane Regimens
Brief Title: A Study of ABT-751 in Patients With Recurrent Breast Cancer After Taxane (Taxol or Taxotere) Therapy.
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Abbott (Industry)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: M02-447
Record Dates: First submitted 2003-06-19; First posted 2003-06-23 (Estimated); Last update posted 2007-11-29 (Estimated); Status verified 2007-11

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — ABT751

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: ABT-751

SUMMARY:
The purpose of the study is to determine if ABT-751 will decrease tumors, and determine how long the tumor shrinkage can be maintained in patients with breast cancer after having had taxol or taxotere. Patients will receive ABT-751 by mouth daily for 21 days. Patients will be off drug for 7 days before starting the next cycle of drug.

ELIGIBILITY:
Inclusion Criteria

* Stage IIIB or IV breast cancer.
* Recurrent tumor after or while on taxane therapy (taxol or taxotere).
* Able to tolerate normal activities of daily living.
* Adequate bone marrow, kidney and liver function.

Exclusion Criteria

* Pregnant or breast feeding.
* No anti-tumor therapy (including hormonal therapy or Herceptin) within 4 weeks of the start of ABT-751 administration.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 40
Dates: Start 2002-11; Study Completion 2004-08 (Actual)

PRIMARY OUTCOMES:
Objective Response Rate in subjects with Breast cancer | 1 year

SECONDARY OUTCOMES:
Time to Tumor Progression (TTP) | 1 year
Survival | 2 years
Toxicities associated with treatment administration | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Helen Eliopoulos, MD, Study Director — Abbott
Locations (8):
- United States (8):
  - Oncology-Hematology Group of South Florida, Miami, Florida
  - Clinical Research Network, Inc., Plantation, Florida
  - Georgia Cancer Specialists, Atlanta, Georgia
  - Northwestern University Medical School Division of Hematology/Oncology, Chicago, Illinois
  - Indiana University Cancer Center Section of of Hemtology/Oncology Indiana Cancer Pavilion, Indianapolis, Indiana
  - Northern Indiana Cancer Research Consortium, South Bend, Indiana
  - Oncology & Hemotology Associates of Kansas City, PA, Kansas City, Missouri
  - Texas Oncology, Dallas, Texas